CLINICAL TRIAL: NCT03892811
Title: Evaluation of the Effect of Flow Rate on Swallowing Function in Young Infants
Status: Withdrawn | Type: Observational
Why Stopped: IRB protocol was not approved by Boston Children's Hospital
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Stephanie DiPerna, AP - Medical Staff, Radiology - Diagnostic, Boston Children's Hospital
Other Study IDs: IRB-P00028852
Record Dates: First submitted 2019-02-06; First posted 2019-03-27 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Deglutition Disorders in Infants; Bottle Feeding
MeSH Terms: conditions — Bottle Feeding

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants referred for swallow study: This is a within-subjects intervention study where each infant in the study will receive all three conditions.
  The three study conditions are bottle-feeding with 1) Dr. Brown's Ultra-Preemie bottle nipple, 2) Dr. Brown's Preemie bottle nipple, and 3) Dr. Brown's Level 1 bottle nipple.
  Interventions: Other: Three study conditions

INTERVENTIONS:
Other: Three study conditions — Continuous fluoroscopy (at 30 frames/second) will be used for intermittent periods to capture 10 swallows in the initial sucking sequence of each of three study conditions: 1) Dr. Brown's Ultra-Preemie bottle nipple, 2) Dr. Brown's Preemie bottle nipple, and 3) Dr. Brown's Level 1 bottle nipple.

SUMMARY:
The purpose of this study is to evaluate the effect of nipple flow rate on swallowing function in infants less than 3 months corrected age (up to 11 weeks and 6 days) who have been referred for videofluoroscopic swallow study.

DETAILED DESCRIPTION:
Feeding difficulties are common in infants born premature and with medical complexity, particularly those with congenital heart disease. One of the most common strategies for managing feeding difficulties is changing the milk flow rate of the bottle nipple. Milk flow is the rate at which milk transfers from the bottle to the infant's mouth. During swallowing, the vocal folds must close to prevent aspiration of fluid into the airway. When milk flow is fast, the infant must swallow frequently to clear the bolus of fluid and prevent aspiration; this is done at the expense of respiration. When the milk flow rate is slowed, the infant can swallow less frequently, allowing better integration of respiration, and has more time to coordinate an effective swallow. While there is some very limited evidence that slower milk flow rate improves feeding in infants born premature and with congenital heart disease, the underlying mechanisms for improvement of feeding remain unknown. This project will be the first to evaluate the effect of milk flow rate on swallowing function under fluoroscopy to better understanding how swallowing changes under different conditions of flow in young infants. This research will provide the evidence needed to support the use of this simple intervention (i.e., changing the flow rate) in infants at risk for feeding difficulty and swallowing dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Infant less than 3 months corrected age
* Must be referred for video fluoroscopic swallow study (VFSS) at Boston Children's Hospital

Exclusion Criteria:

- Infant unsafe to trial all study conditions as determined by clinician(s) conducting the VFSS.

Ages: 12 Hours to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants less than 3 months corrected age (up to 11 weeks and 6 days) who have been referred for video fluoroscopic swallow study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
VFSS - number of sucks per swallow | Through completion of 10 swallows under each study condition, maximum of 1 minute per study condition.
  Number of sucks per swallow for each of 10 swallows under each of the three study conditions.
VFSS - oral bolus control | Through completion of 10 swallows under each study condition, maximum of 1 minute per study condition.
  Oral bolus control for each of 10 swallows under each of the three study conditions.
VFSS - location of swallow onset | Through completion of 10 swallows under each study condition, maximum of 1 minute per study condition.
  Location of swallow onset for each of 10 swallows under each of the three study conditions.
VFSS - presence of pharyngonasal regurgitation | Through completion of 10 swallows under each study condition, maximum of 1 minute per study condition.
  Presence of pharyngonasal regurgitation for each of 10 swallows under each of the three study conditions.
VFSS - presence of laryngeal penetration | Through completion of 10 swallows under each study condition, maximum of 1 minute per study condition.
  Presence of laryngeal penetration for each of 10 swallows under each of the three study conditions.
VFSS - presence of aspiration (silent or non-silent) | Through completion of 10 swallows under each study condition, maximum of 1 minute per study condition.
  Presence of aspiration (silent or non-silent) for each of 10 swallows under each of the three study conditions.
VFSS - presence of post-swallow residue | Through completion of 10 swallows under each study condition, maximum of 1 minute per study condition.
  Presence of post-swallow residue for each of 10 swallows under each of the three study conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A DiPerna, MD, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available in a secure Database.
Time Frame: Data will be made available 2 years after study completion.
Access Criteria: Data access requests will be reviewed by the research team.

REFERENCES:
- [Background] Pados BF, Park J, Dodrill P. Know the Flow: Milk Flow Rates From Bottle Nipples Used in the Hospital and After Discharge. Adv Neonatal Care. 2019 Feb;19(1):32-41. doi: 10.1097/ANC.0000000000000538. PMID 30028734
- [Background] Pados BF, Thoyre SM, Estrem HH, Park J, Knafl GJ, Nix B. Effects of milk flow on the physiological and behavioural responses to feeding in an infant with hypoplastic left heart syndrome. Cardiol Young. 2017 Jan;27(1):139-153. doi: 10.1017/S1047951116000251. Epub 2016 Mar 16. PMID 26982280